CLINICAL TRIAL: NCT00065910
Title: A Joint Attention Intervention With Caregivers and Their Children With Autism
Brief Title: Improving Attention Skills of Children With Autism
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R21MH064927 (NIH)
Record Dates: First submitted 2003-08-01; First posted 2003-08-05 (Estimated); Last update posted 2007-07-02 (Estimated); Status verified 2003-06

CONDITIONS: Autism
Keywords: Joint attention; Developmental delay; Caregiver interaction
MeSH Terms: conditions — Autistic Disorder; Learning Disabilities

INTERVENTIONS:
Behavioral: Caregiver joint attention intervention

SUMMARY:
Toddlers with autism have poor joint attention skills. Joint attention skills include pointing to objects, following another person's gaze, and responding to invitations to join in a social interaction. Improved joint attention skills may lead to better verbal ability as the child ages. This study teaches caregivers how to help their toddlers with autism develop joint attention skills.

DETAILED DESCRIPTION:
Young children with autism show impairment in joint attention. The impairment affects their ability to sustain a shared interest in social interaction and to use specific joint attention skills, such as pointing and showing. The importance of joint attention is underscored by data suggesting these skills are important to later language skills. Targeting joint attention deficits in developmentally young children using familiar caregivers may result in better child language outcomes. This study will teach caregivers how to initiate and maintain episodes of joint engagement with their children.

Participants will be randomized to either the intervention group or to a wait list control group. Each caregiver and child in the intervention group will participate in 24 1-hour sessions, 3 times a week for 8 weeks. In these sessions, caregivers will be taught 10 different modules for teaching joint attention skills to their children. Outcome measures will include language and joint attention skills in the child and caregiver adherence to the intervention protocols. Children and caregivers will be assessed at baseline, during the course of the 8-week intervention, and 10 weeks after the end of the intervention. Participants assigned to the wait list group will begin the intervention at Week 12.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of autism based on Autism Diagnostic Interview-Revised (ADI-R) and Autism Diagnostic Observation Schedule (ADOS) criteria

Exclusion Criteria

* Seizures
* Medical or psychiatric diagnoses other than autism that potentially contribute to developmental delay (e.g., genetic syndromes)

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30
Dates: Start 2001-09; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Connie Kasari, PhD, Principal Investigator — University of California, Los Angelos
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Derived] Kasari C, Gulsrud AC, Wong C, Kwon S, Locke J. Randomized controlled caregiver mediated joint engagement intervention for toddlers with autism. J Autism Dev Disord. 2010 Sep;40(9):1045-56. doi: 10.1007/s10803-010-0955-5. PMID 20145986